CLINICAL TRIAL: NCT00023621
Title: A Phase II Randomized, Double-Blind, Placebo-Controlled Clinical Trial of Celecoxib in Subjects With Basal Cell Nevus Syndrome
Brief Title: Celecoxib in Preventing Basal Cell Carcinoma in Patients With Basal Cell Nevus Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: UCSF-U19-CA81888-BC; CDR0000068817 (Registry Identifier: PDQ (Physician Data Query)); UCSF-H473-16531-02B; NCI-P01-0190
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2007-07

CONDITIONS: Non-melanomatous Skin Cancer
Keywords: basal cell carcinoma of the skin
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Celecoxib

INTERVENTIONS:
Drug: celecoxib

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development of cancer. The use of celecoxib may be an effective way to prevent the development of basal cell carcinoma.

PURPOSE: Randomized phase II trial to determine the effectiveness of celecoxib in preventing basal cell carcinoma in patients who have basal cell nevus syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether celecoxib prevents the development of basal cell carcinoma in patients with basal cell nevus syndrome.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are randomized to 1 of 2 arms.

* Arm I: Patients receive oral celecoxib twice daily.
* Arm II: Patients receive oral placebo twice daily. Treatment continues for 2 years in the absence of unacceptable toxicity.

Patients are followed every 3 months for 3 years.

PROJECTED ACCRUAL: A total of 60 patients (30 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed basal cell carcinoma (BCC)

  * At least 5 prior BCCs AND
  * At least 4 BCCs within the past year
* Meets diagnostic criteria for basal cell nevus syndrome (BCNS)

  * Any 1 of the following:

    * More than 2 BCCs or 1 before age 20
    * Histologically confirmed odontogenic keratocysts of the jaw
    * 3 or more palmar and/or plantar pits
    * Bilamellar calcification of the falx cerebri (if less than 20 years of age)
    * Fused, bifid, or markedly splayed ribs
    * First degree relative with BCNS
    * PTC gene mutation in normal tissue OR
  * Any 2 of the following:

    * Macrocephaly determined after adjustment for height
    * Congenital malformations (e.g., cleft lip or palate, frontal bossing, "coarse face", or moderate or severe hypertelorism)
    * Skeletal abnormalities (e.g., Sprengel deformity, marked pectus deformity, or marked syndactyly of the digits)
    * Radiological abnormalities (e.g., bridging of the sella turcica, vertebral anomalies, modeling defects of the hands and feet, or flame-shaped lucencies of the hands or feet)
    * Ovarian fibroma
    * Medulloblastoma

PATIENT CHARACTERISTICS:

Age:

* 18 to 75

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 3,000/mm^3
* Platelet count greater than 125,000/mm^3
* Hemoglobin greater than 12.0 g/dL (women)
* Hemoglobin greater than 13.0 g/dL (men)
* No significant coagulation defect

Hepatic:

* Bilirubin normal
* ALT/AST no greater than 1.5 times upper limit of normal (ULN)
* No chronic or acute hepatic disorder

Renal:

* Creatinine no greater than 1.5 times ULN
* BUN normal
* Electrolytes within normal
* No chronic or acute renal disorder

Cardiovascular:

* No congestive heart failure

Gastrointestinal:

* No active gastrointestinal disease
* No inflammatory bowel disease
* No chronic or acute pancreatic disorder
* No history of gastrointestinal ulceration allowed except with permission of primary care physician
* No esophageal, gastric, pyloric channel, or duodenal ulceration within the past 30 days
* Stool hematest normal

Other:

* No prior invasive malignancy within the past 5 years except nonmelanoma skin cancer, stage I cervical cancer, stage 0 chronic lymphoblastic leukemia, or medulloblastoma
* No hypersensitivity to COX-2 inhibitors, nonsteroidal anti-inflammatory drugs (NSAIDs), salicylates, or sulfonamides
* No other condition that would preclude study involvement
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 2 weeks since prior topical agents as chemoprevention
* At least 1 year since other prior chemotherapy

Endocrine therapy:

* At least 1 month since prior oral or IV corticosteroids
* At least 6 months since prior inhaled corticosteroid use for longer than 4 weeks
* At least 2 weeks since prior topical glucocorticoids
* No concurrent topical glucocorticoids
* Concurrent oral and IV corticosteroid use of less than 2 weeks within 6 months allowed
* Concurrent inhaled corticosteroid use of less than 4 weeks within 6 months allowed

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* At least 2 weeks since prior topical retinoids or alpha-hydroxy acids (e.g., glycolic acid or lactic acid)
* At least 2 weeks since prior topical medications
* At least 30 days since prior investigational agents
* At least 2 months since prior NSAIDs given more than 3 times/week
* At least 2 months since prior aspirin dose of more than 100 mg/day given more than 3 times/week
* At least 6 months since prior oral retinoids
* No concurrent chronic NSAIDs (more than 3 times per week for at least 2 weeks)
* No concurrent aspirin dose of more than 100 mg/day
* No concurrent topical medications
* No concurrent fluconazole
* No concurrent lithium
* No concurrent retinoids (including topical administration) or alpha-hydroxy acids
* No other concurrent investigational agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2001-02; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Prevention of the development of basal cell carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Ervin Epstein, MD, Study Chair — University of California, San Francisco
Locations (2):
- United States (2):
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York

REFERENCES:
- [Result] Tang JY, Wu A, Linos E, Parimi N, Lee W, Aszterbaum M, Asgari MM, Bickers DR, Epstein EH Jr. High prevalence of vitamin D deficiency in patients with basal cell nevus syndrome. Arch Dermatol. 2010 Oct;146(10):1105-10. doi: 10.1001/archdermatol.2010.247. PMID 20956641